CLINICAL TRIAL: NCT03445455
Title: Assessment of Tidal Volume by Electrical Impendance Tomography During Non Invasive Oxygenation Techniques in de Novo Hypoxemic Acute Respiratory Failure
Brief Title: Assessment of Tidal Volume During Non Invasive Oxygenation Techniques
Acronym: VOLHYPOX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Dr Guillaume CARTEAUX, Associate Professor, Henri Mondor University Hospital
Other Study IDs: 2017-A03560-53
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Failure With Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- De novo AHRF: Acute hypoxemic non hypercapnic respiratory failure with a PaO2/FiO2 ratio < 200.
  The following oxygenation devices are used and assessed during routine care:
  High concentration mask, High flow nasal canula, NIV using buco-nasal mask or Helmet.
  Electro impedence tomography signal will be recorded throughout this assessement for tidal volume measurement
  Interventions: Device: Tidal volume measurement

INTERVENTIONS:
Device: Tidal volume measurement — Recording of thoracic impendance variations during different non-invasive oxygenation techniques.
  Conversion to Tidal volume after calibration using the airway flow signal recorded during the NIV with bucco-nasal mask.

SUMMARY:
High Tidal volume is one of the main mechanisms that lead to lung injuries under mechanical ventilation (ventilator induced lung injury: VILI). It could also induce lung damage during spontaneous or assisted ventilation (patient-self inflicted lung injury: P-SILI). Different non invasive oxygenation devices are available to deliver oxygen during acute hypoxemic respiratory failure: high concentration mask, high flow nasal canula and non-invasive ventilation (with bucco-nasal mask or helmet). The investigators hypothesized that the device may influence the tidal volume. Therefore, the objective of this study is to measure and compare the tidal volume during the use of each device. Tidal volume will be measured using Electrical impedence tomography.

DETAILED DESCRIPTION:
Background : De novo acute respiratory failure with moderate to severe hypoxemia is associated with high intubation and mortality rates. Under non-invasive ventilation (NIV) with a bucco-nasal mask, a high Tidal volume is associated with NIV failure and poor outcome. It is suspected that non-control of the Tidal volume may worsen the prognosis of the patient. Indeed, it is logical to consider that the physiopathological mechanisms that lead to ventilator induced lung injury (VILI) under mechanical ventilation, especially over-distension, can in the same way aggravate pulmonary lesions under NIV and even during spontaneous breathing. The value of the Tidal volume is available in non-invasive ventilation with the bucco-nasal mask, but it is unknown with the use of other non-invasive oxygenation techniques : oxygen therapy with the high concentration mask, non-invasive ventilation with the helmet, and high flow nasal canula.

Objectives : The main objective is to compare the Tidal volume received under different oxygenation techniques (oxygen therapy with high concentration mask, NIV with bucco-nasal mask and with helmet, high flow nasal canula), in patients with de novo acute hypoxemic respiratory failure and moderate to severe hypoxemia.

Methods : All patients admitted in intensive care for de novo acute hypoxemic respiratory failure, non hypercapnic, with moderate to severe hypoxemia (PiO2/FiO2 < 200 mmHg) will be included. Patients with one of the following items will be excluded : chronic respiratory disease, cardiogenic pulmonary edema, hemodynamic instability, coma, contraindication to NIV, indication for immediate intubation.

After inclusion, the Tidal volume will be measured for each technique with the use of electrical impedance tomography, in a random order. Randomisation will be carried out by using sealed envelopes containing a predetermined order. Each technique will be used for 15 minutes. For NIV with the bucco-nasal mask, the inspiratory pressure will be progressively adjusted to maintain the Tidal volume between 6 and 8 ml/kg of ideal body weight without dropping below 7 cm H2O and the positive expiratory pressure will be gradually increased to 5 cm H2O. For NIV with the helmet, the inspiratory pressure will be progressively increase to 12 cm H2O and the positive expiratory pressure will be gradually increased to 5 cm H2O. For high flow nasal canula,the gas flow will be set at 50 L/minute. FiO2 will be adjusted to keep SpO2 above 92%. To convert the thoracic impedance variations into absolute values of Tidal volumes, the airway flow signal will be collected with a pneumotacograph during the NIV with bucco-nasal mask session. The following data will also be collected : respiratory rate, comfort, regional Tidal volume in dependent and non-dependent areas and global inhomogeneity index, Pa02, PaCO2 and pH (If an arterial catheter is present). Signed consent will be required prior to any inclusion.

Expected benefits : This study will provide a better understanding of P-Sili and help define the place each non-invasive oxygenation techniques in the management of de novo acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory rate > 25 per minute
* PaO2/FiO2 < 200 mmHg
* PaCO2 < 45 mmHg
* Signed consent by patient or relative

Exclusion Criteria:

* Chronic respiratory disease
* COPD exacerbation
* Acute asthma
* Cardiogenic pulmonary edema
* Hemodynamic instability (systolic blood pressure < 90 mmHg or mean blood pressure < 65 mmHg or use of catecholamines)
* Coma (Glasgow coma scale < 12)
* Contraindication to non-invasive ventilation
* Indication to immediate intubation according to the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with de novo acute hypoxemic respiratory failure
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Tidal volume | Averaged value over the last 3 minutes of thoracic impedance recording
  in milliliter

SECONDARY OUTCOMES:
pH | After 15 minutes of using a non invasive oxygenation device
  Arterial blood gases will be collected only if an arterial catheter will be already inserted
PaO2 | After 15 minutes of using a non invasive oxygenation device
  in mm Hg; Arterial blood gases will be collected only if an arterial catheter will be already inserted
PaCO2 | After 15 minutes of using a non invasive oxygenation device
  in mm Hg; Arterial blood gases will be collected only if an arterial catheter will be already inserted
Respiratory rate | After 15 minutes of using a non invasive oxygenation device
  in cycle/min
Comfort | After 15 minutes of using a non invasive oxygenation device
  using a semiquantitative scale from 1 (the worst comfort) to 5 (the best comfort)
Regional Tidal volume | Averaged value over the last 3 minutes of thoracic impedance recording
  in milliliter
Global inhomogeneity index | Averaged value over the last 3 minutes of thoracic impedance recording
  in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Carteaux, MD, PhD, Principal Investigator — Henri Mondor University Hospital